CLINICAL TRIAL: NCT05005455
Title: A Randomized, Double-blind, Parallel Controlled, Single-dose Phase I Clinical Study to Evaluate Pharmacokinetic Similarity, Safety, and Immunogenicity of Bevacizumab With Different Manufacturing Process in Healthy Male Subjects
Brief Title: Study of Bevacizumab With Different Manufacturing Process in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CIBI305K101
Record Dates: First submitted 2021-07-17; First posted 2021-08-13 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Healthy Male Subjects
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bevacizumab with old manufacturing process. (Active Comparator)
  Interventions: Drug: bevacizumab with old manufacturing process.
- bevacizumab with new manufacturing process. (Experimental)
  Interventions: Drug: bevacizumab with new manufacturing process.

INTERVENTIONS:
Drug: bevacizumab with new manufacturing process. — 3mg/kg,I.V.,single dose
  Arms: bevacizumab with new manufacturing process.
Drug: bevacizumab with old manufacturing process. — 3mg/kg,I.V.,single dose
  Arms: bevacizumab with old manufacturing process.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic similarity of bevacizumab with different manufacturing process in healthy male subjects. Another purpose is to determine safety, and immunogenicity of bevacizumab with different manufacturing process.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form and fully understand the test content, process and possible adverse reactions, and be able to complete the study according to the test plan requirements;
* Age≥18 years and ≤50 years, healthy male subjects;
* Weight ≥ 50kg and ≤ 100kg,BMI≥ 19kg/m2 and < 28 kg/m2
* Clinical examinations in the screening period are normal or abnormal without clinical significance.
* Agree to take effective contraceptive measures throughout the study period and until at least 6 months after receiving the last dose of study drug

Exclusion Criteria:

1. Any prior VEGF(vascular endothelial growth factor) and VEGFR(Vascular Endothelial Growth Factor Receptor) antibody or protein treatment within one year.
2. Serious, non-healing wound, active ulcer, or untreated bone fracture, or major surgical procedure within 2 months prior to randomization or anticipation of need for major surgery during the course of the study or 2 months after end of the study.
3. Use Rx or OTC drugs or nutritional health products within 5 half-lives or within 2 weeks before the first dose of study drug (According to the longer time).Herbal supplements need to stop at 28 days before the first dose of study drug.
4. Positive hepatitis b surface antigen (HBsAg), hepatitis c virus (HCV) antibody, or human immunodeficiency virus (HIV) antibody or syphilis.
5. Known hypersensitivity to bevacizumab or any excipients, known allergic disease or allergic constitution.
6. History of blood donation within 3 months before the first dose of study drug.
7. Treatment with any other investigational agent or participation in another clinical trial within 3 months prior to screening.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Age≥18 years and ≤50 years, healthy male subjects
Enrollment: 100 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure:Area Under the Curve(AUC0-∞) | 84days

SECONDARY OUTCOMES:
Area Under the Curve(AUClast) | 84days
Maximum Concentration (Cmax) | 84days
Volume of distribution (V) | 84days
Total body clearance (CL) | 84days
Elimination half-life (t1/2) | 84days
Time at which maximum concentration occurred (Tmax) | 2016days
Incicende of Adverse Events (AEs) | 98days
Anti-drug Antibody（ADA）and Neutralizing Antibody（NAb） | 98days

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of Soochow university, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No